CLINICAL TRIAL: NCT06017687
Title: Data Collection and Evaluation of a Mobile, Machine-learning-based Solution for Blood Pressure Estimation - the OptiBP Study.
Brief Title: Data Collection and Evaluation of OptiBP Under Investigational Use
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biospectal (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: US Data Collection Study
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: General Population

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Principal Arm (Other): Each participant will use the OptiBP Study app on their smartphone
  Interventions: Device: OptiBP Study app

INTERVENTIONS:
Device: OptiBP Study app — Each participant will use OptiBP Study app to measure their blood pressure optically by applying their fingertip to their smartphone camera, and subsequently enter the blood pressure values obtained by measuring it with their own blood pressure cuff.

SUMMARY:
The purpose of this study is to collect data to develop and evaluate the use of state-of-the-art machine learning approaches within a mobile phone application for the estimation of blood pressure.

DETAILED DESCRIPTION:
Participants will simultaneously acquire blood pressure measurements through a cuff-based, automatic, over-the-counter blood pressure monitor on the upper arm, while recording an optical signal through the camera of a smartphone on the tip of the index of the opposite arm.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years old (at least 19 years old in Alabama and Nebraska, at least 21 years old in Puerto Rico);
2. Live in the United States of America
3. Have an Android smartphone
4. Have access to an arm-worn blood pressure monitor (cuff)
5. Have access to the Google Play store to download the OptiBP study app on their phone
6. Be comfortable communicating in written and spoken English
7. Be willing and able to provide informed consent to participate in the study

Exclusion Criteria:

1. Known contact dermatitis to nickel/chromium
2. Lesion or deficiency on hand, preventing placing a finger on the smartphone camera
3. Known dysrhythmia like bigeminy, trigeminy, isolated VPB, atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500000 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Collect Blood Pressure (BP) data and assess performance of smartphone based BP estimations models | 12 months
  To collect data to train a machine-learning based solution for estimating blood pressure. Participants will simultaneously acquire blood pressure measurements through a cuff-based, automatic, over-the-counter blood pressure monitor at the upper arm, while recording an optical signal through the camera of a smartphone on the tip of the index of the opposite arm. The performance of the machine learning model will be assessed by calculating the mean and standard deviation of the error of blood pressure estimations versus cuff-based, automatic, over-the-counter blood pressure monitors.

SECONDARY OUTCOMES:
Safety by assessing inconvenience and adverse events | 12 months
  To identify potential use errors of an app that use the machine-learning model to estimate blood pressure. And to assess safety of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Frappereau, Principal Investigator — Biospectal
Locations (1):
- Decentralized Trial, Truckee, California, United States

IPD SHARING:
Plan to Share IPD: No
The data is anonymized and used for machine learning training